CLINICAL TRIAL: NCT06779149
Title: Efficacy of CBT-I and Lemborexant Medication for Different Subtypes of Chronic Insomnia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Toronto Metropolitan University (Other); The Royal Ottawa Mental Health Centre (Other)
Responsible Party: Principal Investigator, Charles M. Morin, Professor, Laval University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-3057
Record Dates: First submitted 2025-01-12; First posted 2025-01-16 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Insomnia Disorder
Keywords: Insomnia; Cognitive behavioral therapy for insomnia; Lemborexant; Insomnia phenotypes; Objective short sleep duration
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — lemborexant

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Participants assigned to the medication groups (active and placebo) and their prescribing physicians will be blind to medication treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cognitive Behavioral Treatment for Insomnia (CBT-I) (Experimental): Participants in this treatment group will receive CBT-I. CBT-I sessions will occur weekly for the first 4 sessions and biweekly for the last 2 sessions (treatment phase is thus 8 weeks). : Graduate level students in clinical psychology will serve as therapists for this project.
  Interventions: Behavioral: Cognitive Behavioral Treatment for Insomnia (CBT-I)
- Lemborexant medication (Experimental): Participants assigned to this group will be prescribed 5 to 10 mg of lemborexant to be taken at bedtime in 5 mg capsules. Lemborexant (Dayvigo) is a Dual Orexin Receptor Antagonist approved by Health Canada for the treatment of adult with insomnia, characterized by difficulties with sleep onset and/or sleep maintenance. Pharmacy staff will package medications for each participant in a generic bottle labeled with the participant's ID code and treatment dates (identical for the lemborexant and placebo arms). Six consultation visits will be conducted during the 8-week treatment phase to monitor treatment response and drug side effects. The starting dose will be 5 mg with titration to 10 mg if needed (i.e., based on clinical response and tolerability) following the first week.
  Interventions: Drug: Lemborexant
- Placebo (Placebo Comparator): Participants assigned to this group will be prescribed 5 to 10 mg of placebo to be taken at bedtime in 5 mg capsules identical to lemborexant. Pharmacy staff will package medications for each participant in a generic bottle labeled with the participant's ID code and treatment dates (identical for the lemborexant and placebo arms). Six consultation visits will be conducted during the 8-week treatment phase to monitor treatment response and drug side effects. The starting dose will be 5 mg with titration to 10 mg if needed (i.e., based on clinical response and tolerability) following the first week.
  Interventions: Drug: Placebo

INTERVENTIONS:
Behavioral: Cognitive Behavioral Treatment for Insomnia (CBT-I) — Participants in this treatment group will receive CBT-I. CBT-I sessions will occur weekly for the first 4 sessions and biweekly for the last 2 sessions (treatment phase is thus 8 weeks). : Graduate level students in clinical psychology will serve as therapists for this project.
  Arms: Cognitive Behavioral Treatment for Insomnia (CBT-I)
Drug: Lemborexant — Participants assigned to this group will be prescribed 5 to 10 mg of lemborexant to be taken at bedtime in 5 mg capsules. Lemborexant (Dayvigo) is a Dual Orexin Receptor Antagonist approved by Health Canada for the treatment of adult with insomnia, characterized by difficulties with sleep onset and/or sleep maintenance. Pharmacy staff will package medications for each participant in a generic bottle labeled with the participant's ID code and treatment dates (identical for the lemborexant and placebo arms). Six consultation visits will be conducted during the 8-week treatment phase to monitor treatment response and drug side effects. The starting dose will be 5 mg with titration to 10 mg if needed (i.e., based on clinical response and tolerability) following the first week.
  Arms: Lemborexant medication
Drug: Placebo — Participants assigned to this group will be prescribed 5 to 10 mg of placebo to be taken at bedtime in 5 mg capsules identical to lemborexant. Pharmacy staff will package medications for each participant in a generic bottle labeled with the participant's ID code and treatment dates (identical for the lemborexant and placebo arms). Six consultation visits will be conducted during the 8-week treatment phase to monitor treatment response and drug side effects. The starting dose will be 5 mg with titration to 10 mg if needed (i.e., based on clinical response and tolerability) following the first week.
  Arms: Placebo

SUMMARY:
The primary aims of this study is to contrast the effectiveness of CBT-I and pharmacotherapy (lemborexant) compared to placebo on sleep and mental health outcomes in people with insomnia disorder and anxiety/depressive symptoms. In addition, the study will evaluate whether insomnia phenotypes (i.e., +/- 6hrs of sleep) at baseline moderate the effectiveness of the intervention on both sleep and mental health outcomes.

DETAILED DESCRIPTION:
Participants meeting study criteria will be randomized to one of three conditions (1:1:1) involving a 8-week treatment protocol (6 consultations over an 8-week period): 1) CBT-I, 2) an active hypnotic medication (lemborexant, 5-10 mg at bedtime) or 3) a placebo medication. A stratified-based variable block randomization schedule will be used to assign eligible patients to study arms once they have completed baseline measures. Stratification will be based on objective (EEG-defined) sleep duration (< 6 h vs. > 6 h) and age (< 50 years old vs. > 50 years old).

CBT-I will be provided in six therapy sessions provided over an 8-week period by trained graduate therapists in clinical psychology. Lemborexant and placebo medication (compounded and coded by a pharmacy) will be provided by consulting physicians (blinded) in six consultations over an 8-week period. Physicians will have the option of increasing the initial starting dose from 5 mg to 10 mg if needed. Control participants will receive a placebo medication identical in size and color to the active medication.

The assessment phase will include baseline, post-treatment, and 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older at the time of enrolment
* Meeting Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria for insomnia disorder (Duke Sleep Interview), with total Insomnia Severity Index (ISI) score > 10, and score ≥ 2 on either the interference or distress item
* Minimal symptoms of anxiety and/or depression with Patient Health Questionnaire (PHQ-9) > 4 and/or Generalized Anxiety Disorder (GAD-7) > 4
* Ability to read and understand French or English
* Ability to use a smartphone, tablet, or computer, and access to home internet connection

Exclusion Criteria:

* Presence of a lifetime diagnosis of any psychotic or bipolar disorder
* Untreated psychiatric disorder (e.g., major depression) or risk for suicide
* Substance/alcohol use disorder within the past year
* Any life-threatening or progressive medical illness (e.g., cancer, chronic obstructive pulmonary disease) or neurological degenerative disease (e.g., dementia)
* Current use of sleep-promoting medications (prescribed or over-the-counter) or cannabis-derived products for sleep more than two nights per week
* Current use of tricyclic antidepressants, monoamine oxidase inhibitors, or atypical antidepressants
* Reported diagnosis of sleep disorder other than insomnia (e.g., obstructive sleep apnea, restless legs syndrome, rapid eye movement behavior disorder, delayed phase sleep disorder, narcolepsy)
* Total score > 5 on the Stop-Bang Questionnaire and/or clinical symptoms suggestive of sleep apnea (excessive daytime sleepiness), or Epworth score > 10, restless legs syndrome or other signs of other sleep disorders
* Atypical sleep schedules (i.e., habitual bedtimes later than 2:00 AM and rising times later than 10:00 AM on more than two days/nights per week as documented from a sleep diary)
* Working night shifts more than five nights per month in the last six months
* Consuming 2 or more alcoholic beverages per day regularly (3 days or more per week)
* Any contra-indications to using the study medication, including lung disease/breathing problems (e.g., chronic obstructive pulmonary disease), use of strong or moderate CYP3A inducers (strong - rifampin, carbamazepine, and St. John's Wort) (moderate - bosentan, efavirenz, etravirine, and modafinil), pregnant and breastfeeding women
* Not using any method of birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Insomnia Symptom Severity | Baseline, during treatment period (weeks 0-8), at the end of the 2-week post-treatment and 6-month follow-up.
  Insomnia symptoms will be measured by the Insomnia Severity Index (ISI). The ISI is a self-report questionnaire evaluating seven dimensions of insomnia-severity of sleep onset, sleep maintenance, early morning awakening problems, sleep dissatisfaction, interference of sleep difficulties with daytime functioning, noticeability of sleep problems by others, and distress caused by sleep difficulties. Each item is rated on a 0 to 4 scale and the total score ranges from 0 to 28, with a higher total score suggesting more severe insomnia symptoms. An ISI score < 8 will be used to define remission. Treatment response will be defined at each assessment as a reduction of 8 points or more on the ISI compared with the baseline score.

SECONDARY OUTCOMES:
Sleep onset latency from sleep diary | Nightly during 2-week pre-treatment, treatment period (weeks 0-8), 2-week post-treatment and 6-month follow-up.
  Mean sleep onset latency per night in minutes from sleep diary.
Wake after sleep onset from sleep diary | Nightly during 2-week pre-treatment, treatment period (weeks 0-8), 2-week post-treatment and 6-month follow-up.
  Mean wake after sleep onset per night in minutes from sleep diary.
Total sleep time from sleep diary | Nightly during 2-week pre-treatment, treatment period (weeks 0-8), 2-week post-treatment and 6-month follow-up.
  Mean total sleep time per night in minutes from sleep diary.
Sleep efficiency from sleep diary | Nightly during 2-week pre-treatment, treatment period (weeks 0-8), 2-week post-treatment and 6-month follow-up.
  Mean sleep efficiency per night in percentage from sleep diary.
Depressive symptoms | Baseline, at the end of the 2-week post-treatment and 6-month follow-up.
  The presence of symptoms of depression will be assessed by the Patient Health Questionnaire-9 (PHQ-9). Scores range from 0 to 27, with scores of 15 and higher suggesting the need for treatment.
Anxiety symptoms | Baseline, at the end of the 2-week post-treatment and 6-month follow-up.
  Anxiety symptom severity will be measured by the Generalised Anxiety Disorder 7-item (GAD-7). Scores range from 0 to 21, with scores of 15 and over suggesting severe anxiety.
Mental well-being | Baseline, at the end of the 2-week post-treatment and 6-month follow-up.
  Mental well-being will be measured by the 5-item World Health Organisation Well-Being Index (WHO-5). Scores range from 0 to 100, with higher scores indicating higher well-being.
Fatigue | Baseline, at the end of the 2-week post-treatment and 6-month follow-up.
  Fatigue severity will be measured by the 9-item Fatigue Severity Scale (FSS). Scores range from 9 to 63 . higher score indicates more severe fatigue and impairment.
Functional impact of insomnia | Baseline, at the end of the 2-week post-treatment and 6-month follow-up.
  Work and Social Adjustment Scale (WSAS) of 5 items will be used to measure how much sleep issues impair ability to function in terms of work, home management, leisure, and relationships. Scores range from 0 to 40. Higher scores indicate more work and social impairment.
Sleep-related beliefs and attitudes | Baseline, at the end of the 2-week post-treatment and 6-month follow-up.
  Sleep-related beliefs and attitudes will be measured by the Dysfunctional Beliefs and Attitudes about Sleep (DBAS-16). Higher scores indicate more dysfunctional beliefs and attitudes about sleep. The total score is calculated from the average score of all the items on the scale and could range from 0 to 10.

OTHER OUTCOMES:
Cognitive performance | Baseline and at the end of the 2-week post-treatment.
  Changes in cognitive performance measured by Cognitive Failures Questionnaire 2.0 (CFQ 2.0) will serve as an exploratory outcome. The CFQ 2.0 is a 15-item questionnaire asking respondents to rate the frequency with which they make minor mistakes (e.g., forgetting to take their keys, calling people by the wrong name). Scores range from 0 to 60, with higher scores indicating greater frequency of cognitive failures.

CONTACTS AND LOCATIONS:
Overall Officials: Charles M Morin, PhD, Principal Investigator — Université Laval Centre d'étude des troubles du sommeil
Locations (1):
- Université Laval Centre d'étude des troubles du sommeil, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen SJ, Ivers H, Dang-Vu TT, Shapiro CM, Carney CE, Robillard R, Morin CM. Efficacy of cognitive behavioral therapy for insomnia and lemborexant medication for different subtypes of chronic insomnia: study protocol for a randomized controlled trial. BMC Psychiatry. 2025 May 9;25(1):470. doi: 10.1186/s12888-025-06878-1. PMID 40346496